CLINICAL TRIAL: NCT03948399
Title: The Prevalence of a Low Ankle-Brachial Index in Patients With Acute Cerebral Ischemic Event.
Brief Title: The Prevalence of a Low Ankle-Brachial Index in Acute Cerebral Ischemia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jan Biziel University Hospital No 2 in Bydgoszcz (Other)
Responsible Party: Principal Investigator, Pawel Sokal, Paweł Sokal, Jan Biziel University Hospital No 2 in Bydgoszcz
Other Study IDs: JBUH-ABI-CIE-2018
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; TIA; ABI; LEAD
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STROKE GROUP: 150 patients admitted to Stroke Unit with a diagnosis of acute ischemic stroke (IS) or transient ischemic attack (TIA)
  Interventions: Device: Duplex scanning of carotid arteries; Device: ABI measurement
- CONTROL GROUP: 50 individuals admitted to hospital without diagnosis of acute cerebrovascular disease; with diagnosis of dizziness, epilepsy, sclerosis multiplex.
  Interventions: Device: Duplex scanning of carotid arteries; Device: ABI measurement

INTERVENTIONS:
Device: Duplex scanning of carotid arteries — Measurement of carotid arteries
Device: ABI measurement — ankle brachial index (ABI) assessment

SUMMARY:
Aim of the study is assessment the prevalence of the low ankle-brachial index (ABI) defined less than or equal 0.9 in patients with acute cerebral ischemic event (stroke or transient ischemic attack) and determinate the correlation between ABI and internal carotid artery stenosis (ICAS) in the acute cerebral ischemic patients.

The low ABI is a strong marker of generalized atherosclerosis. LEAD is a strong independent predictor for stroke.

DETAILED DESCRIPTION:
Aim of the study is assessment the prevalence of the low ankle-brachial index (ABI) defined less than or equal 0.9 in patients with acute cerebral ischemic event (stroke or transient ischemic attack) and determinate the correlation between ABI and internal carotid artery stenosis (ICAS) in the acute cerebral ischemic patients.

The ABI is a non-invasive tool useful for the diagnosis of LEAD. The low ABI is a strong marker of generalized atherosclerosis. LEAD is a strong independent predictor for stroke. Significant ICAS is prevalent among patients having LEAD. Acute ischemic stroke due to significant ICAS has poor prognosis.

Patients with LEAD may be a suitable subgroup for screening for ICAS using duplex scanning.

Estimating the relationship between cerebral ischemic event and the ABI value could help better guide preventive and risk reduction strategies.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke or transient ischemic attack of anterior circulation
* Consent of patient

Exclusion Criteria:

* primary intracranial hemorrhage,
* venous sinus thrombosis,
* unconsciousness,
* intubation,
* inability to provide and write a consent application form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending to hospital settings diagnosed with acute ischemic event (stroke or TIA) and control group individuals undergo computed tomography (CT) or magnetic resonance imaging (MRI) of the brain, lipid profile, had stroke risk factors assessed.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
ABI | 7 days
  Prevalence of a low ankle-brachial index (ABI) in patients with acute cerebral ischemic event

SECONDARY OUTCOMES:
ABI/ICAS | 7 days
  Correlation between ABI and internal carotid artery stenosis (ICAS) in the acute cerebral ischemic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Sokal, Ph.D., Principal Investigator — Jan Biziel University Hospital Collegium Medicum Nicolaus Copernicus University
Locations (1):
- Department of Neurosurgery and Neurology University Hospital nr 2 Collegium Medicum Nicolaus Copernicus University, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No